CLINICAL TRIAL: NCT06120894
Title: Strip Meniscometry in Dry Eye Evaluation in Connection With Cataract Surgery
Brief Title: Strip Meniscometry in Dry Eye Evaluation
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Zuzana Schreiberova, Principal Investigator, University Hospital Olomouc
Other Study IDs: 24/22
Record Dates: First submitted 2023-11-01; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye; Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Tonometry, Ocular; Slit Lamp Microscopy; Refraction, Ocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Central visual acuity — Measurement of central visual acuity using Snellen optotype chart.
Diagnostic Test: Intraocular pressure measurement — Measurement of intraocular pressure using non-contact Canon TX-20P tonometer.
Diagnostic Test: Slit lamp examination — Slit lamp examination of the anterior and posterior segment of the eye after pharmacological dilation of the pupil using application of short-time mydriatics (1% tropicamide and 10% phenylephrine).
Diagnostic Test: Refraction and keratometry — Measurement of refraction and keratometry using refractometer Nidek ARK-1a.
Diagnostic Test: Optical biometry — Measurement of optical biometry using biometer Argos (Barrett or SRK/T formula).
Diagnostic Test: Strip meniscometry (SM) — Strip meniscometry examination using strip meniscometry tube.
Diagnostic Test: Lid Parallel Conjunctival Folds test (LIPCOF) — Evaluation of lid parallel conjunctival folds using slit lamp examination.
Diagnostic Test: Staining of the ocular surface with fluorescein — Evaluation of ocular surface fluorescein staining using Oxford scheme.
Diagnostic Test: Tear break up time test (TBUT) — Evaluation of tear break up time using slit lamp examination.
Other: Ocular Surface Disease Index questionnaire (OSDI) — Evaluation of Ocular Surface Disease Index using Ocular Surface Disease Index questionnaire.

SUMMARY:
Strip meniscometry is a relatively new method for evaluating the tear meniscus. The aim of the study is to evaluate the possible effect of cataract surgery on ocular surface disease and to assess the possible benefit of strip meniscometry in the preoperative and postoperative evaluation of patients.

DETAILED DESCRIPTION:
Cataract surgery is one of the most successful anterior segment surgeries and usually results in excellent postoperative visual acuity. However, some patients may experience symptoms of dry eye disease after a successful procedure, most commonly a foreign body sensation in the eye, intermittent pain, and blurred vision. These problems then interfere with normal daily activities and also reduce the patient's satisfaction with the surgery.

The new method for tear film examination Strip meniscometry (SM) appears to be a suitable alternative to the Schirmer test. SM values correlate with Oxford score (fluorescein staining), tear break up time test or measurement of meniscus height using anterior segment optical coherence tomography. It is a minimally invasive and rapid examination method that measures the volume of the aqueous component of the tear film.

The aim of this study is to evaluate the possible influence of cataract surgery on the development of iatrogenic OSD and to assess the contribution of a new diagnostic method, SM, for the evaluation of OSD before and after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* performing of pre-operative examination before cataract surgery
* signed informed consent

Exclusion Criteria:

* use of antiglaucoma drugs
* chronic blepharitis
* previous viral keratitis
* previous keratoplasty or laser refractive surgery
* known systemic disease causing changes on ocular surface (diabetes mellitus, connective tissue disease)
* use of medication causing changes on ocular surface (antidepressant, beta blockers)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group will be recruited from patients who undergo cataract surgery at the Department of Ophthalmology of University Hospital Olomouc and Palacky University.
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in strip meniscometry. | Week 1, 4, 12
  Strip Meniscometry Tube in millimeters.

SECONDARY OUTCOMES:
Change in ocular surface fluorescein staining. | Week 1, 4, 12
  Oxford scheme grading with range from 0 (none staining dots) to 5 (severe dry eye).
Change in tear film stability. | Week 1, 4, 12
  Tear break up time test in seconds.
Change in lid-parallel conjunctival folds evaluation. | Week 1, 4, 12
  Lid-parallel conjunctival folds (LIPCOF) grading from 0 (no conjunctival folds) to 3 (more than two permanent and clear parallel folds (normally higher than 0.2 mm).
Change in Ocular Surface Disease Index. | Week 1, 4, 12
  Ocular Surface Disease Index (OSDI) questionnaire with range from 0 to 100 (higher score represents greater disability).

CONTACTS AND LOCATIONS:
Overall Officials: Marta Karhanova, MD, PhD, Principal Investigator — University Hospital Olomouc and Palacky University Olomouc
Locations (1):
- Department of Ophthalmology, University Hospital Olomouc, Olomouc, Czechia